CLINICAL TRIAL: NCT00443404
Title: Double Blind, Placebo Controlled Study for the Study of the Effectiveness of Perioperative Analgesia in Phantom and Stump Pain
Brief Title: Optimized Perioperative Analgesia Reduces the Prevalence and the Intensity of Phantom Pain in Lower Limb Amputation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Diamanto Aretha, University Hospital of Patras
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: phantom pain-UPatras; There are no secondary Id
Record Dates: First submitted 2007-03-05; First posted 2007-03-06 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2009-09

CONDITIONS: Phantom Limb Pain
Keywords: phantom; amputation; analgesia; pain; preemptive; perioperative; lower limb amputation; intensity of phantom limb pain; preemptive analgesia reduces phantom pain; perioperative analgesia reduces phantom pain; Severe Phantom Limb Pain (VAS>70 mm); resistant to medical treatment one week before amputation
MeSH Terms: conditions — Phantom Limb; Agnosia; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Active Comparator): perioperative epidural analgesia
  Interventions: Procedure: perioperative epidural catheter
- 2 (Active Comparator): Iv PCA Fentanyl preoperative, Epidural analgesia postoperative
  Interventions: Procedure: perioperative epidural catheter
- 3 (Active Comparator): perioperative IV PCA Fentanyl, epidural anesthesia
  Interventions: Procedure: perioperative epidural catheter
- 4 (Active Comparator): perioperative IV PCA Fentanyl general anesthesia
  Interventions: Procedure: perioperative epidural catheter
- 5 (Placebo Comparator): IV PCA with saline 0.9% and sc saline 0.9%in the L3-L4 area. IM meperidine, po codeine/acetaminophen, IV acetaminophen and IV parecoxib
  Interventions: Procedure: perioperative epidural catheter

INTERVENTIONS:
Procedure: perioperative epidural catheter — Perioperative epidural catheter in groups 1-4. Pre- and postoperative epidural analgesia in group 1. Preoperative IV PCA Fentanyl and postoperative epidural analgesia in group 2. Perioperative IV PCA Fentanyl in groups 2,3. IM meperidine p.o. codeine/acetaminophen, IV acetaminophen and IV parecoxib in group 5 (control)

SUMMARY:
Severe pre-amputation pain is associated with phantom pain development, and phantom pain models assign major importance to central and peripheral nervous system changes related to pre-amputation pain. Several interventions have been evaluated for phantom pain prevention, including continuous brachial plexus blockade5, intravenous6 or epidural ketamine administration, postoperative perineural ketamine/clonidine infusion8 and oral gabapentin9, but their true effect remains unclear.

DETAILED DESCRIPTION:
In a prospective, randomized, double-blind trial, 65 patients undergoing elective lower limb amputation were assigned to one of five analgesic regimens. Patients in groups 1-4 had lumbar epidural catheter placed 48 hours before amputation, and received epidural bupivacaine/fentanyl or saline infusion before and/or after amputation. Patients receiving epidural saline also had IV Fentanyl Patient-Control Analgesia, whereas patients receiving epidural analgesia also had IV saline. Group 5 (control) received IM meperidine and oral codeine/acetaminophen. VAS and McGill Pain Questionnaire (MPQ) scores (for ischemic, phantom and stump pain) were recorded starting 48 hours before, continuing until 48 hours after amputation, and at 4 days, 10 days, 1 and 6 months after amputation. Phantom and stump pain intensity and frequency were the main study endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age >18, Visual Analog. Scale (VAS) pain score >70mm which was frequent or continuous one week before scheduled major (above or below knee) amputation, and patient consent.

Exclusion Criteria:

* No written patient consent
* Age < 18 years
* Age > 82 years
* Antiplatelet medication
* Mental status not acceptable
* Exclusion criteria were age >85
* Emergency amputation
* Ipsilateral re-amputation
* Foot or toe amputation
* Inability to complete a detailed pain questionnaire
* History of chronic pain or substance abuse
* Active psychiatric disease requiring treatment
* Any contraindication to epidural catheter placement (anticoagulation, anti-platelet medications, previous lumbar spine surgery).

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-12; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
VAS and McGill PRI(R)2 scores for phantom and stump pain are recorded 48 and 24 hours before, and 4 and 10 days, 1 and 6 months after amputation. Phantom and stump pain intensity are the endpoints of the study. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Diamanto N. Aretha, MD, Principal Investigator — University of Patras, School of Medicine, University Hospital of Patras, Rion, 26500, Department of Anaesthesiology and Critical Care Medicine; Menelaos Karanikolas, MD, MPH, Study Director — University of Patras, School of Medicine, University Hospital of Patras, Rion, 26500, Department of Anaesthesiology and Critical Care Medicine; Kriton S Filos, MD Professor, Study Chair — University of Patras, School of Medicine, University Hospital of Patras, Rion, 26500, Department of Anaesthesiology and Critical Care Medicine; Georgia Monantera, MD, Principal Investigator — University of Patras, School of Medicine, University Hospital of Patras, Rion, 26500, Department of Anaesthesiology and Critical Care Medicine; Ioannis Tsolakis, MD Professor, Study Director — University of Patras, School of Medicine, University Hospital of Patras, Rion, 26500, Department of Surgery
Locations (1):
- Pátrai, Greece

REFERENCES:
- [Derived] Karanikolas M, Aretha D, Tsolakis I, Monantera G, Kiekkas P, Papadoulas S, Swarm RA, Filos KS. Optimized perioperative analgesia reduces chronic phantom limb pain intensity, prevalence, and frequency: a prospective, randomized, clinical trial. Anesthesiology. 2011 May;114(5):1144-54. doi: 10.1097/ALN.0b013e31820fc7d2. PMID 21368651